CLINICAL TRIAL: NCT03224793
Title: A Blinded, Safety, Tolerability, and Pharmacokinetic Study of Single Doses of BIIB059 in Healthy Japanese Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of Single Doses of BIIB059 in Healthy Japanese Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 230HV101
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BIIB059 20 mg (Experimental): Participants will receive single subcutaneous (SC) dose of 20 milligram (mg) BIIB059 or matching placebo on Day 1.
  Interventions: Drug: BIIB059; Drug: Placebo
- BIIB059 50mg (Experimental): Participants will receive single SC dose of 50 mg BIIB059 or matching placebo on Day 1.
  Interventions: Drug: BIIB059; Drug: Placebo
- BIIB059 150mg (Experimental): Participants will receive single SC dose of 150 mg BIIB059 or matching placebo on Day 1.
  Interventions: Drug: BIIB059; Drug: Placebo
- BIIB059 450mg (Experimental): Participants will receive single SC dose of 450 mg BIIB059 or matching placebo on Day 1.
  Interventions: Drug: BIIB059; Drug: Placebo

INTERVENTIONS:
Drug: BIIB059 — Administered as specified in the treatment arm
Drug: Placebo — Administered as specified in the treatment arm

SUMMARY:
To assess the safety and tolerability of single, subcutaneous (SC) doses of BIIB059 in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations
* Must have been born in Japan, and both their biological parents and grandparents must have been of Japanese origin
* Aged 18 to 55 years old, inclusive, at the time of informed consent, and must have a body mass index between 18 and 30 kilogram per square meter (kg/m2), and a body weight >45 kg
* All women of childbearing potential and all men must practice highly effective contraception during the study and for 16 weeks after their dose of study treatment

Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator
* History or positive test result for human immunodeficiency virus. Current active hepatitis C virus infection (defined as hepatitis C virus RNA above the limit of detection). Positive test result for hepatitis B virus (defined as positive for hepatitis B surface antigen or hepatitis B core antibody). Chronic, recurrent, or serious infection (e.g., pneumonia, septicemia), as determined by the Investigator, within 90 days prior to Screening or between Screening and Day -1
* Clinically significant abnormal laboratory test values, as determined by the Investigator, at Screening or Day -1
* Current enrollment or a plan to enroll in any interventional clinical study in which an investigational treatment or approved therapy for investigational use is administered within 5 half-lives prior to Day -1
* History of alcohol or substance abuse (as determined by the Investigator), a positive urine drug or alcohol test at Screening or Day -1, an unwillingness to refrain from illicit or recreational drugs, or an unwillingness to abide by the alcohol restrictions

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 20 weeks
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose: results in death; life-threatening event; requires inpatient hospitalization; significant disability; congenital anomaly; medically important event.
Percentage of Participants With Clinically Significant Abnormal Clinical Laboratory Parameters, Vital Signs, 12-Lead Electrocardiograms (ECG), and Physical Examination Findings | Up to 20 weeks
Percentage of Participants With Anti-BIIB059 Antibodies | Up to 20 weeks

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve From Time 0 to 28 Days Post-dose (AUC0-28d) | Up to 28 days
Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Measurable Concentration (AUClast) | Up to 112 days
Maximum Observed Concentration (Cmax) | Up to 112 days
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf), | Up to 112 days
Time to Reach Maximum Observed Concentration (Tmax) | Up to 112 days
Terminal Half-Life (t1/2) | Up to 112 days
Time of Last Measurable Concentration (Tlast) | Up to 112 days
Apparent Total Clearance (CL/F) | Up to 112 days
Apparent Volume of Distribution (Vz/F) | Up to 112 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States